CLINICAL TRIAL: NCT02604433
Title: A Phase 3, Double-Blind, Placebo Controlled Multicenter Study to Determine the Efficacy and Safety of Luspatercept (ACE-536) in Adults With Transfusion Dependent Beta (B)-Thalassemia
Brief Title: An Efficacy and Safety Study of Luspatercept (ACE-536) Versus Placebo in Adults Who Require Regular Red Blood Cell Transfusions Due to Beta (β) Thalassemia
Acronym: BELIEVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACE-536-B-THAL-001
Record Dates: First submitted 2015-10-21; First posted 2015-11-13 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Erythrocyte Transfusion; Beta-Thalassemia
Keywords: ACE-536; Safety; Efficacy; Placebo; Red Blood Cell Transfusions; Beta -Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Luspatercept (ACE-536) plus Best Supportive Care (BSC) (Experimental): Luspatercept, subcutaneous(ly) (SC) once every 21 days
  Interventions: Drug: Luspatercept
- Placebo plus Best Supportive Care (BSC) (Placebo Comparator): normal saline solution subcutaneous(ly) (SC) once every 21 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Luspatercept — Subjects will start with luspatercept at 1 mg/kg dose level.
  Other Names: ACE-536
  Arms: Luspatercept (ACE-536) plus Best Supportive Care (BSC)
Other: Placebo — Placebo, Subcutaneous, every 21 days.
  Arms: Placebo plus Best Supportive Care (BSC)

SUMMARY:
This is a Phase 3, double-blind, randomized, placebo-controlled, multicenter study to determine the efficacy and safety of luspatercept (ACE-536) plus Best supportive care (BSC) versus placebo plus BSC in adults who require regular red blood cell transfusion due to (β)-thalassemia.

The study is divided into the following periods:

* Historical Period,
* Screening/Run-in Period,
* Double-blind Treatment Period (48 weeks),
* Double-blind Long-term Treatment Period, (at the investigator's discretion an additional 48 weeks),
* Open-Label Phase post unblinding and upon Data Monitoring Committee positive recommendation
* Post-treatment Follow-up Period

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Male or female, ≥18 years of age at the time of signing the informed consent document (ICF).
2. Subject must understand and voluntarily sign an Inform Consent Form prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Documented diagnosis of β-thalassemia or Hemoglobin E/β-thalassemia. (β-thalassemia with mutation and/or multiplication of alpha globin is allowed).
5. Regularly transfused, defined as: 6-20 Red Blood Cell (RBC) units* in the 24 weeks prior to randomization and no transfusion-free period for ≥ 35 days during that period.

   * Sites who prescribe transfusions and have the transfusion records only in volumes should use for conversion of volume to units the below criteria, in order to obtain number of units within the last 24 weeks to assess the eligibility: 1 unit in this protocol refers to a quantity of packed RBCs approximately 200-350 mL. (i) sites who use transfusion bags within this range, or ≥ 350 mL, the conversion in units should be done by dividing the volume transfused to the patient by 350 mL, (ii) sites who use transfusion bags < 200 mL, the conversion in units should be done by dividing the volume transfused to the patient by 200 mL.
6. Performance status: Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
7. A female of childbearing potential (FCBP) for this study is defined as a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months). FCBP participating in the study must:

   1. Have two negative pregnancy tests as verified by the Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence ** from heterosexual contact.
   2. Either commit to true abstinence** from heterosexual contact (which must be reviewed on a monthly basis and source documented) If a FCBP engages in sexual activity that may result in a pregnancy, she must agree to use, and be able to comply with, effective*** contraception without interruption, 28 days prior to starting investigational product, during the study therapy (including dose interruptions), and for 12 weeks (approximately five times the mean terminal half-life of luspatercept based on multiple-dose Pharmacokinetic PK) data) after discontinuation of study therapy.

      * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.] *** Agreement to use highly effective methods of contraception that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly throughout the course of the study.

   Such methods include: Combined (estrogen and progesterone/progestin containing) hormonal contraception: Oral; Intravaginal; Transdermal; Progestogen/progestin only hormonal contraception associated with inhibition of ovulation: Oral; Injectable hormonal contraception; Implantable hormonal contraception; Placement of an intrauterine device (IUD); Placement of an intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomized partner; Sexual Abstinence.
8. Male subjects must:

   * Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks (approximately five times the mean terminal half-life of luspatercept based on multiple-dose PK data) following investigational product discontinuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. A diagnosis of Hemoglobin S/β-thalassemia or alpha (α)-thalassemia (eg, Hemoglobin H);
5. Evidence of active hepatitis C (HCV) infection as demonstrated by a positive HCV-RNA test of sufficient sensitivity, or active infectious hepatitis B as demonstrated by the presence of HBsAg and/or HBVDNA-positive,, or known positive human immunodeficiency virus (HIV).

   Note: Subjects receiving antiviral therapies should have 2 negative HCVRNA tests 3 months apart.(ie, one test at the end of the antiviral therapy and a second test 3 months following the first test).
6. Deep Vein Thrombosis (DVT) or stroke requiring medical intervention ≤ 24 weeks prior to randomization.
7. Use of chronic anticoagulant therapy is excluded, unless the treatment stopped at least 28 days prior to randomization. Anticoagulant therapies used for prophylaxis for surgery or high risk procedures as well as low Molecular Weight (LMW) heparin for superficial venous thrombosis and chronic aspirin are allowed.
8. Platelet count > 1000 x 109/L
9. Poorly controlled diabetes mellitus within 24 weeks prior to randomization as defined by short term (eg, hyperosmolar or ketoacidotic crisis) and/or history of diabetic cardiovascular complications (eg, stroke or myocardial infarction).
10. Treatment with another investigational drug or device ≤ 28 days prior to randomization.
11. Prior exposure to sotatercept (ACE-011) or luspatercept (ACE-536).
12. Use of an erythropoiesis-stimulating agent (ESA) ≤ 24 weeks prior to randomization.
13. Iron chelation therapy, if initiated ≤ 24 weeks prior to randomization (allowed if initiated > 24 weeks before or during treatment).
14. Hydroxyurea treatment ≤ 24 weeks prior to randomization.
15. Pregnant or lactating females.
16. Uncontrolled hypertension. Controlled hypertension for this protocol is considered ≤ Grade 1 according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (current active minor version).
17. Major organ damage, including:

    1. Liver disease with alanine aminotransferase (ALT) > 3 x the upper limit of normal (ULN) or history of evidence of cirrhosis;
    2. Heart disease, heart failure as classified by the New York Heart Association (NYHA) classification 3 or higher, or significant arrhythmia requiring treatment, or recent myocardial infarction within 6 months of randomization.
    3. Lung disease, including pulmonary fibrosis or pulmonary hypertension which are clinically significant ie, ≥ Grade 3 NCI CTCAE version 4.0 (current active minor version).
    4. Creatinine clearance < 60 mL/min (per Cockroft-Gault formula).
18. Proteinuria ≥ Grade 3 according to NCI CTCAE version 4.0 (current active minor version).
19. Chronic systemic glucocorticoids ≤ 12 weeks prior to randomization (physiologic replacement therapy for adrenal insufficiency is allowed). Single day glucocorticoid treatment (eg, for prevention or treatment of transfusion reactions, is allowed).
20. Major surgery ≤ 12 weeks prior to randomization (subjects must have completely recovered from any previous surgery prior to randomization).
21. History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product (see Investigator Brochure).
22. Cytotoxic agents, immunosuppressants ≤ 28 days prior to randomization (ie, antithymocite globulin (ATG) or cyclosporine)
23. History of malignancy with the exception of:

    1. Curatively resected nonmelanoma skin cancer.
    2. Curatively treated cervical carcinoma in situ.
    3. Other solid tumor with no known active disease in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (76):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Australia (6):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital Institute of Medical and Veterinary Science, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Prince Alfred Hospital, Camperdown
- Bulgaria (3):
  - University Mulitiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Specialized Hospital for Active Treatment of Haematological Diseases - Sofia, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Marina EAD, Varna
- University Health Network, Toronto, Ontario, Canada
- France (4):
  - Hopital Henri Mondor, Créteil
  - GH de Institut Catholique St. VincentHématologie, Lille
  - Hopitaux de La Timone, Marseille
  - Hospital of Necker, Paris
- Greece (7):
  - Laiko General Hospital of Athens, Ampelokipi - Athens
  - Local Institution - 405, Ampelokipi - Athens
  - General Children's Hospital "Agia Sophia", Athens
  - General Hospital Georgios Gennimatas of Athens, Athens
  - University General Hospital of Patras, Rio Patras
  - Hippokration Hospital, Thessaloniki
  - Local Institution - 404, Thessaloniki
- Israel (7):
  - Soroka University Medical Centre, Beersheba
  - Rambam Health Corporation, Haifa
  - HaEmek Medical Center, Haïfa (Afula)
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
- Italy (10):
  - Presidio Ospedaliero Antonio Perrino, Brindisi
  - Universita degli Studi di Cagliari - ASL8, Cagliari
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Ferrara
  - Ente Ospedaliero Ospedali Galliera - Centro della Microcitemia e delle Anemie Congenite, Genoa
  - Fondazione Ca Granda IRCCS Ospedale Maggiore, Milan
  - Seconda Universita Degli Studi Di Napoli, Naples
  - AORN A Cardarelli, Napoli
  - Azienda Ospedaliero Universitaria S. Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Chronic Care Center, Beirut, Lebanon
- Malaysia (7):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Pulau Pinang c/o Penang Medical College, George Town
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
- Thailand (3):
  - Chulalongkorn University Faculty of Medicine - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Chiang Mai University - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Tunisia (4):
  - University Hospital Farhat Hached, Sousse
  - Bone Marrow Transplant Center, Tunis
  - Aziza Othmana Hospital, Tunis
  - Military Hospital of Tunis, Tunis
- Turkey (Türkiye) (8):
  - Acibadem Adana Hospital, Adana
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Local Institution - 524, Adana
  - Hacettepe Universitesi, Ankara
  - Antalya Egitim Arastirma, Antalya
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Mersin University Medical Faculty, Mersin
- United Kingdom (5):
  - St James University Hospital, Leeds
  - Barts Health NHS Trust - The Royal London Hospital, London
  - Whittington Hospital, London
  - University College Hospital Trust, London Bloomsbury
  - Manchester Royal Infirmary, Manchester

REFERENCES:
- [Result] Porter J. Beyond transfusion therapy: new therapies in thalassemia including drugs, alternate donor transplant, and gene therapy. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):361-370. doi: 10.1182/asheducation-2018.1.361. PMID 30504333
- [Result] Piga A, Perrotta S, Gamberini MR, Voskaridou E, Melpignano A, Filosa A, Caruso V, Pietrangelo A, Longo F, Tartaglione I, Borgna-Pignatti C, Zhang X, Laadem A, Sherman ML, Attie KM. Luspatercept improves hemoglobin levels and blood transfusion requirements in a study of patients with beta-thalassemia. Blood. 2019 Mar 21;133(12):1279-1289. doi: 10.1182/blood-2018-10-879247. Epub 2019 Jan 7. PMID 30617198
- [Derived] Cappellini MD, Viprakasit V, Georgiev P, Coates TD, Origa R, Khelif A, Liew HK, Tantiworawit A, Chew LP, Khalil A, Ho PJ, Kuo KHM, Holot N, Perin M, Giuseppi AC, Kuo WL, Lai Y, Medlin LF, Bueno LM, Kattamis A, Taher AT. Long-term efficacy and safety of luspatercept for the treatment of anaemia in patients with transfusion-dependent beta-thalassaemia (BELIEVE): final results from a phase 3 randomised trial. Lancet Haematol. 2025 Mar;12(3):e180-e189. doi: 10.1016/S2352-3026(24)00376-4. Epub 2025 Feb 10. PMID 39947215
- [Derived] Garbowski MW, Ugidos M, Risueno A, Shetty JK, Schwickart M, Hermine O, Porter JB, Thakurta A, Vodala S. Luspatercept stimulates erythropoiesis, increases iron utilization, and redistributes body iron in transfusion-dependent thalassemia. Am J Hematol. 2024 Feb;99(2):182-192. doi: 10.1002/ajh.27102. Epub 2023 Oct 2. PMID 37782758
- [Derived] Denton CC, Vodala S, Veluswamy S, Hofstra TC, Coates TD, Wood JC. Splenic iron decreases without change in volume or liver parameters during luspatercept therapy. Blood. 2023 Nov 30;142(22):1932-1934. doi: 10.1182/blood.2023021839. PMID 37704579
- [Derived] Cappellini MD, Taher AT. The use of luspatercept for thalassemia in adults. Blood Adv. 2021 Jan 12;5(1):326-333. doi: 10.1182/bloodadvances.2020002725. PMID 33570654
- [Derived] Cappellini MD, Viprakasit V, Taher AT, Georgiev P, Kuo KHM, Coates T, Voskaridou E, Liew HK, Pazgal-Kobrowski I, Forni GL, Perrotta S, Khelif A, Lal A, Kattamis A, Vlachaki E, Origa R, Aydinok Y, Bejaoui M, Ho PJ, Chew LP, Bee PC, Lim SM, Lu MY, Tantiworawit A, Ganeva P, Gercheva L, Shah F, Neufeld EJ, Thompson A, Laadem A, Shetty JK, Zou J, Zhang J, Miteva D, Zinger T, Linde PG, Sherman ML, Hermine O, Porter J, Piga A; BELIEVE Investigators. A Phase 3 Trial of Luspatercept in Patients with Transfusion-Dependent beta-Thalassemia. N Engl J Med. 2020 Mar 26;382(13):1219-1231. doi: 10.1056/NEJMoa1910182. PMID 32212518
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 336 participants were randomized, 332 participants were treated.
Groups:
- Luspatercept + BSC: Luspatercept (ACE-536) was administered subcutaneously (SC) at a starting dose level of 1 mg/kg once every 21 days. Participants could be dose-titrated to 1.25 mg/kg, but the maximum total dose should not exceed 120 mg, total dose per administration during the Treatment Period, the Long-term Treatment Period, and Open-Label Treatment Period. BSC = Best Supportive Care
- Placebo + BSC: Placebo (normal saline) was administered subcutaneously (SC) in volumes to match active treatment once every 21 days. BSC = Best Supportive Care
Period: Overall Study
Arm/Group | Luspatercept + BSC | Placebo + BSC
Started (Participants randomized) | 224 | 112
Participants Treated (All participants who received at least 1 dose of study drug) | 223 | 109
Completed 24 Weeks of Treatment | 211 | 102
Completed 48 Weeks of Treatment | 202 | 96
Completed 96 Weeks of Treatment | 155 | 3
Completed 144 Weeks of Treatment | 125 | 0
Completed 192 Weeks of Treatment | 6 | 0
Completed (Completed study per original protocol) | 6 | 6
Not Completed | 218 | 106
Not completed — Withdrawal by Subject | 37 | 16
Not completed — Adverse Event | 4 | 0
Not completed — Other reasons | 3 | 5
Not completed — Death | 4 | 1
Not completed — Transition to Rollover Protocol | 169 | 82
Not completed — Physician Decision | 1 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Luspatercept + BSC | Placebo + BSC | Total
Number analyzed (Participants) | 224 | 112 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (10.67) | 31.9 (9.89) | 32.1 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 63 | 195
  Male | 92 | 49 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 218 | 107 | 325
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 81 | 36 | 117
  Black or African American | 1 | 0 | 1
  White | 122 | 60 | 182
  Not collected or reported | 5 | 5 | 10
  Other | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Erythroid Response - Week 13 to Week 24
Description: Erythroid Response was defined as red blood cell (RBC) transfusion burden reduction from baseline ≥ 33% with a reduction of at least 2 units during Week 13 - 24 compared to the 12-week interval on or prior to Dose 1 Day 1.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Weeks 13 to Week 24
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 224 | 112
Percentage of participants | 21.0 | 4.5
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Odds ratio 95% confidence intervals (CIs), and p-value were estimated from the Cochran Mantel-Haenszel (CMH) test stratified by the geographical regions defined at randomization; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Significance level of 0.050 for 2-sided tests; Odds Ratio (OR) = 5.62, 95% CI 2-sided [2.17 to 14.53]
Statistical Analysis 2: Comparison: Luspatercept + BSC vs Placebo + BSC; Test type: Superiority; Difference in Percentages = 16.5, 95% CI 2-sided [10.0 to 23.1] — Luspatercept - Placebo
Statistical Analysis 3: Comparison: Luspatercept + BSC vs Placebo + BSC; Test type: Superiority; Common Risk Difference = 16.5, 95% CI [9.9 to 23.1] — Luspatercept - Placebo

2. Secondary Outcome: Percentage Of Participants Who Achieved ≥ 33% Reduction From Baseline in Transfusion Burden - Week 37 to Week 48
Description: Percentage of participants who achieved a red blood cell (RBC) transfusion burden reduction from baseline ≥ 33% with a reduction of at least 2 units during Weeks 37 - 48 compared to the 12-week interval on or prior to Dose 1 Day 1.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Weeks 37 to Week 48
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 224 | 112
Percentage of participants | 19.6 | 3.6
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Odds ratio 95% CIs, and p-value were estimated from the CMH test stratified by the geographical regions defined at randomization. To control the overall Type 1 error rate for outcomes 2-4, the testing procedure was implemented strictly in order: the test for this outcome was only conducted when there was evidence showing that erythroid response was achieved in the luspatercept group from Week 13 to Week 24 (primary endpoint); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Significance level of 0.050 for 2-sided tests; Odds Ratio (OR) = 6.44, 95% CI 2-sided [2.27 to 18.26]

3. Secondary Outcome: Percentage Of Participants Who Achieve ≥ 50% Reduction From Baseline in Transfusion Burden - Week 13 to Week 24
Description: Percentage of participants who achieved a red blood cell (RBC) transfusion burden reduction from baseline ≥ 50% with a reduction of at least 2 units during Weeks 13 - 24 compared to the 12-week interval on or prior to Dose 1 Day 1.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Weeks 13 to Week 24
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 224 | 112
Percentage of participants | 7.1 | 1.8
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Odds ratio, 95% CIs, and p-value were estimated from the Cochran-Mantel-Haenszel (CMH) test stratified by the geographical regions defined at randomization. To control the overall Type 1 error rate, the testing procedure was done strictly in order: the test for this outcome was only conducted when there was evidence showing erythroid response was achieved in the luspatercept group for the primary endpoint, and 33% hematological improvement was achieved in the luspatercept group in outcome 2; Test type: Superiority; p = 0.0402, Cochran-Mantel-Haenszel — Significance level of 0.050 for 2-sided tests; Odds Ratio (OR) = 4.24, 95% CI 2-sided [0.96 to 18.79]

4. Secondary Outcome: Percentage Of Participants Who Achieve ≥ 50% Reduction From Baseline in Transfusion Burden - Week 37 to Week 48
Description: Percentage of participants who achieved a red blood cell (RBC) transfusion burden reduction from baseline ≥ 50% with a reduction of at least 2 units during Week 37 to Week 48 compared to the 12-week interval on or prior to Dose 1 Day 1.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Week 37 to Week 48
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 224 | 112
Percentage of participants | 10.3 | 0.9
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Odds ratio, 95% CIs, and p-value were estimated from the Cochran-Mantel-Haenszel (CMH) test stratified by the geographical regions defined at randomization. To control the overall Type 1 error rate, the testing procedure was done strictly in order: the test for this outcome was only conducted when there was evidence showing erythroid response was achieved in the luspatercept group for the primary endpoint, and achievement of objective in the luspatercept group in outcomes 2+3; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel — Significance level of 0.050 for 2-sided tests; Odds Ratio (OR) = 11.92, 95% CI 2-sided [1.65 to 86.29]

5. Secondary Outcome: Mean Change From Baseline in Transfusion Burden - Week 13 to Week 24
Description: Baseline was defined as the total number of Red Blood Cells (RBC) units transfused during the 12-week interval on or prior to Dose 1 Day 1. This is compared to the total number of RBC units transfused during the 12-week interval from treatment weeks 13-24.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Weeks 13 to Week 24
Population: All randomized participants with available measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 210 | 102
RBC units | -0.67 (1.792) | 0.66 (1.774)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Change from baseline at Week 48 LSM = least squares mean; Test type: Superiority; p < 0.0001, ANCOVA — Significance level of 0.050 for 2-sided tests; Estimates were based on an ANCOVA model with geographical regions defined at randomization and baseline transfusion burden as covariates; LSM Difference = -1.34, 95% CI 2-sided [-1.76 to -0.93] — luspatercept - placebo

6. Secondary Outcome: Mean Change From Baseline In Liver Iron Concentration (LIC) At Week 48
Description: Baseline was defined as the last value on or before the first dose of study drug was administered; if multiple values were present for the same date, the average of these values was used. If a participant had 1 postbaseline assessment, it was used as the Week 48 value. If a participant had multiple postbaseline assessments, the last one was used as the Week 48 value. The value of LIC was collected by magnetic resonance imaging. Participants with a LIC value > 43 mg/g were not included in the analysis.
Time Frame: Baseline: Week -12 to Day -1; Treatment: Week 48
Population: All randomized participants with available measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 185 | 99
mg/g dry weight | 0.05 (5.770) | -0.00 (5.329)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Change from baseline at Week 48 P-value ANCOVA model with geographical regions defined at randomization and baseline LIC as covariates. LS = least square; Test type: Superiority; p = 0.7598, ANCOVA — Significance level of 0.050 for 2-sided tests; LS Mean of Difference = 0.20, 95% CI 2-sided [-1.10 to 1.51] — luspatercept - placebo

7. Secondary Outcome: Mean Change From Baseline In Mean Daily Dose Of Iron Chelation Therapies (ICT) At Week 48
Description: Three different types of Iron Chelation Therapy (ICT) were analyzed: 1. Deferasirox 2. Deferiprone 3. Deferoxamine Mesilate/Deferoxamine The baseline mean daily dose was calculated using the ICT dosage during the 12 weeks prior to first study drug administration and the postbaseline mean daily dose was calculated during the last 12 weeks of the 48-week double-blind Treatment Period or the last 12 weeks of the study treatment for early discontinued participants.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Week 37 to Week 48
Population: All randomized participants with available measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 129 | 66
mg
  Deferasirox: number analyzed (Participants) | 93 | 49
  Deferasirox | -105.0 (378.67) | -60.4 (297.11)
  Deferiprone: number analyzed (Participants) | 30 | 12
  Deferiprone | -229.1 (893.62) | -73.4 (614.80)
  Deferoxamine Mesilate/Deferoxamine: number analyzed (Participants) | 6 | 5
  Deferoxamine Mesilate/Deferoxamine | 84.9 (523.45) | 274.2 (613.05)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Deferasirox: Change from baseline at Week 48 LS = least squares; Test type: Superiority; p = 0.2552, ANCOVA — Significance level of 0.050 for 2-sided tests; Estimates are based on an ANCOVA model with geographical regions defined at randomization and baseline ICT as covariates; LS Mean of Difference = -68.0, 95% CI 2-sided [-185.8 to 49.7] — luspatercept - placebo
Statistical Analysis 2: Comparison: Luspatercept + BSC vs Placebo + BSC; Deferiprone: Change from baseline at Week 48 LS = least squares; Test type: Superiority; p = 0.7746, ANCOVA — Significance level of 0.050 for 2-sided tests; [statistical method as in outcome 7, analysis 1]; LS Mean of Difference = -76.4, 95% CI 2-sided [-612.9 to 460.1] — luspatercept - placebo
Statistical Analysis 3: Comparison: Luspatercept + BSC vs Placebo + BSC; Deferoxamine Mesilate / Deferoxamine: Change from baseline at Week 48 LS = least squares; Test type: Superiority; p = 0.5186, ANCOVA — Significance level of 0.050 for 2-sided tests; [statistical method as in outcome 7, analysis 1]; LS Mean of Difference = -147.3, 95% CI 2-sided [-673.1 to 378.5] — luspatercept - placebo

8. Secondary Outcome: Mean Change From Baseline In Mean Serum Ferritin At Week 48
Description: For each participant, the baseline mean serum ferritin level was calculated during the 12 weeks prior to first study drug administration. The postbaseline mean serum ferritin level was calculated during the last 12 weeks of the 48-week double-blind Treatment Period or last 12 weeks of study treatment, if discontinued early. The change was calculated as the difference of post baseline mean serum ferritin level and baseline mean serum ferritin level.
Time Frame: Baseline: Day -83 to Day 1; Treatment: Week 37 to Week 48
Population: All randomized participants with available measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 207 | 101
μg/L | -247.19 (713.767) | 100.38 (522.047)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Change from baseline at Week 48 LS = least squares; Test type: Superiority; p < 0.0001, ANCOVA — Significance level of 0.050 for 2-sided tests; Estimates based on an ANCOVA model with geographical regions defined at randomization and baseline serum ferritin as covariates; LS Mean of Difference = -342.59, 95% CI 2-sided [-498.30 to -186.87] — luspatercept - placebo

9. Secondary Outcome: Mean Change From Baseline In Total Hip And Lumbar Spine Bone Mineral Density (BMD) At Week 48
Description: For BMD, the lumbar spine and total hip were measured at baseline and 48 weeks by dual energy x-ray absorptiometry (DXA). Baseline was defined as the last value on or before the first dose of study drug is administered; if multiple values are present for the same date, the average of these values was used. If during the 48 week double-blinded treatment period, a participant has only one assessment, it is counted as 'Week 48' visit; if a participant has multiple assessments, the last one is used as 'Week 48' visit. The analysis was done on the population that had at least 2 measurements.
Time Frame: Baseline: Day 1; Treatment: Week 48
Population: All randomized participants with available measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 190 | 97
gm/cm^2
  Total Hip | 0.01 (0.050) | 0.01 (0.057)
  Lumbar Spine: number analyzed (Participants) | 189 | 97
  Lumbar Spine | -0.00 (0.063) | 0.00 (0.078)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Total Hip Bone Mineral Density: Change from baseline at Week 48 LS = least squares; Test type: Superiority; p = 0.9201, ANCOVA — Significance level of 0.050 for 2-sided tests; Estimates are based on an ANCOVA model with geographical regions defined at randomization and baseline BMD measurement as covariates; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.01 to 0.01] — luspatercept - placebo
Statistical Analysis 2: Comparison: Luspatercept + BSC vs Placebo + BSC; Lumbar Spine Bone Mineral Density: Change from baseline at Week 48 LS = least squares; Test type: Superiority; p = 0.4620, ANCOVA — Significance level of 0.050 for 2-sided tests; [statistical method as in outcome 9, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.02 to 0.01] — luspatercept - placebo

10. Secondary Outcome: Mean Change From Baseline In Myocardial Iron At Week 48
Description: Myocardial Iron levels were measured by Magnetic Resonance Imaging (MRI), using MRI parameter T2* (Unit: ms). T2* values correlates with heart failure (HF) risk (e.g. T2*<6ms: high HF risk).
Time Frame: Baseline: Day 1; Treatment: Week 48
Population: All randomized participants with available measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 201 | 102
ms | -1.83 (15.084) | -0.01 (6.780)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Change from baseline at Week 48 LS = least square; Test type: Superiority; p = 0.0543, ANCOVA — Significance level of 0.050 for 2-sided tests; Estimates were based on an ANCOVA model with geographical regions defined at randomization and baseline myocardial T2* as covariates; LS Mean of Difference = -2.22, 95% CI 2-sided [-4.48 to 0.04] — luspatercept - placebo

11. Secondary Outcome: Mean Change From Baseline in the Transfusion-dependent Quality of Life (TranQol) Questionnaire At Week 24
Description: The TranQol is a self-administered quality of life tool developed for beta-thalassemia patients. The adult self-report version used in this study, includes 36 questions assessed on a 5-point response, that are grouped into 5 domains (Physical Health, Emotional Health, Sexual Health, Family Functioning, School/Career Functioning). Scores are calculated according to specific scoring algorithms developed by the authors. Both individual domains score and the total score range from 0 (worst) to 100 (best). Total Score and Physical Health domain score are reported. Positive change from baseline values indicate improvement.
Time Frame: Baseline: 4 weeks prior to Day 1; Treatment: Week 24
Population: All randomized participants with an evaluable TranQoL questionnaire at screening visit and at least one post-screening visit
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 200 | 94
Score on a scale
  Physical Health Domain Score - Change from Baseline | -1.5 (14.26) | -0.7 (14.24)
  Total Score - Change from Baseline | 0.8 (11.56) | -0.4 (11.62)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Physical Health Domain Score - Change from Baseline at Week 24; Test type: Superiority; p = 0.666, t-test, 2 sided — Significance level of 0.050 for 2-sided tests
Statistical Analysis 2: Comparison: Luspatercept + BSC vs Placebo + BSC; Total Score - Change from Baseline at Week 24; Test type: Superiority; p = 0.384, t-test, 2 sided — Significance level of 0.050 for 2-sided tests

12. Secondary Outcome: Mean Change From Baseline in the 36-item Short Form Health Survey (SF-36) Questionnaire At Weeks 24
Description: The SF-36 (version 2) is a generic, self-administered instrument consisting of 8 multi-item scales that assess 8 health domains. The raw score for each health domain is transformed into a 0 (worst) to 100 (best) domain score. The 0-100 scale score for each health domain is further converted to normbased scores using a T-score transformation, with a mean of 50 and a standard deviation (SD) of 10. Higher norm-based T-scores indicate better heath/QoL. The domains/summaries reported are: 1. Physical Functioning (Range of possible T-scores is 19.26 - 57.54) 2. General Health (Range of possible T-scores is 18.95 - 66.50) 3. Physical Component summary (PCS) (Range of possible T-scores is 5.02 - 79.78). Positive change from baseline values indicate improvement.
Time Frame: Baseline: 4 weeks prior to Day 1; Treatment: Weeks 24
Population: All randomized participants with an evaluable SF-36 questionnaire at screening visit and at least one post-screening visit
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 210 | 103
T-score
  Physical Functioning Domain Score - Change from Baseline: number analyzed (Participants) | 197 | 91
  Physical Functioning Domain Score - Change from Baseline | -0.3 (6.93) | -0.2 (7.86)
  General Health Domain Score - Change from Baseline: number analyzed (Participants) | 197 | 91
  General Health Domain Score - Change from Baseline | 0.4 (7.18) | 0.3 (7.03)
  PCS - Change from Baseline: number analyzed (Participants) | 197 | 91
  PCS - Change from Baseline | -0.4 (7.01) | -0.3 (7.97)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; Physical Functioning Domain - Change from Baseline at Week 24; Test type: Superiority; p = 0.918, t-test, 2 sided — Significance level of 0.050 for 2-sided tests
Statistical Analysis 2: Comparison: Luspatercept + BSC vs Placebo + BSC; General Health Domain - Change from Baseline at Week 24; Test type: Superiority; p = 0.857, t-test, 2 sided — Significance level of 0.050 for 2-sided tests
Statistical Analysis 3: Comparison: Luspatercept + BSC vs Placebo + BSC; PCS - Change from Baseline at Week 24; Test type: Superiority; p = 0.839, t-test, 2 sided — Significance level of 0.050 for 2-sided tests

13. Secondary Outcome: Number of Participants Who Utilized Healthcare Resources During Study
Description: Number of participants who had any of the following types of Healthcare Resource Utilization (HRU): - a doctor office visit (non-study scheduled) - an emergency department visit - a hospitalization
Time Frame: From informed consent signing (up to 12 weeks before start of treatment) to end of treatment (up to approximately 227 weeks)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 224 | 112
Participants
  Doctor Office Visit | 186 | 69
  Emergency Department Visit | 71 | 22
  Hospital Admission | 61 | 5

14. Secondary Outcome: Number of Days Spent in Higher Care Hospital Units
Description: Types of hospitals units considered to be 'higher care' are: - Intensive Care Unit - Coronary Care Unit
Time Frame: as for outcome 13
Population: All randomized participants who spent time in higher care hospital units
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 43 | 5
Days | 8.0 (23.70) | 0.6 (0.55)

15. Secondary Outcome: Percentage Of Participants Who Were Transfusion Independent For ≥ 8 Weeks During Treatment
Description: Transfusion independence was defined as the absence of any transfusion during any consecutive "rolling" 8-week time interval within the treatment period, i.e, Days 1 to 56, Days 2 to 57 and so on.
Time Frame: From first dose through 3 weeks post last dose (up to approximately 218 weeks)
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 224 | 112
Percentage of participants | 12.1 | 1.8
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel — Significance level of 0.050 for 2-sided tests; Odds Ratio (OR) = 7.6, 95% CI 2-sided [1.8 to 32.9]

16. Secondary Outcome: Duration of Reduction in Transfusion Burden
Description: Responders were defined as subjects who achieved ≥ 33% reduction or ≥ 50% reduction in Red Blood Cells Transfusion (RBC-T) burden from baseline with a reduction of at least 2 RBC units during any rolling 12-week interval. The duration of reduction is calculated as Last Day of Response - First day of response +1
Time Frame: From first dose to end of study treatment (up to approximately 215 weeks)
Population: All randomized participants with ≥ 33% reduction or ≥ 50% reduction in RBC-T burden
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 173 | 39
Days
  Number of participants analyzed for 33% | 627.3 (390.54) | 224.0 (155.15)
  Number of participants analyzed for 50%: number analyzed (Participants) | 112 | 9
  Number of participants analyzed for 50% | 491.1 (386.37) | 193.0 (142.51)

17. Secondary Outcome: Longest Duration of Transfusion Independence
Description: Transfusion independence was defined as the absence of any transfusion during any consecutive "rolling" 8-week time interval within the treatment period, ie, Days 1 to 56, Days 2 to 57 and so on. Longest duration of transfusion independence was estimated based on Kaplan-Meier model.
Time Frame: From first dose through 3 weeks post last dose (up to approximately 218 weeks)
Population: All randomized participants who were transfusion independent for ≥ 8 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 27 | 2
Days | 72.0 [62.0 to 103.0] | 71.5 [62.0 to NA] — Insufficient number of events to determine the upper limit

18. Secondary Outcome: Time to Erythroid Response
Description: Time to erythroid response was defined as the time from first dose of the study drug to first erythroid response. This is reported for participants with a ≥ 33% reduction from baseline in RBC transfusion burden (with a reduction of at least 2 units) for any 12-week interval., as well as participants with a ≥ 50% reduction from baseline in RBC transfusion burden (with a reduction of at least 2 units) for any 12-week interval.
Time Frame: From first dose to 48 weeks following first dose
Population: All randomized participants who achieved erythroid response
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 173 | 39
Days
  ≥ 33% Transfusion Burden Reduction | 96.3 (163.92) | 163.5 (148.78)
  ≥ 50% Transfusion Burden Reduction: number analyzed (Participants) | 112 | 9
  ≥ 50% Transfusion Burden Reduction | 189.1 (257.69) | 160.9 (160.17)
Statistical Analysis 1: Comparison: Luspatercept + BSC vs Placebo + BSC; ≥ 33% Transfusion Burden Reduction; Test type: Superiority; p = 0.0195, t-test, 2 sided — Significance level of 0.050 for 2-sided tests; Mean Difference (Final Values) = -67.27, 95% CI 2-sided [-123.63 to -10.91] — luspatercept - placebo
Statistical Analysis 2: Comparison: Luspatercept + BSC vs Placebo + BSC; ≥ 50% Transfusion Burden Reduction; Test type: Superiority; p = 0.7473, t-test, 2 sided — Significance level of 0.050 for 2-sided tests; Mean Difference (Final Values) = 28.24, 95% CI 2-sided [-144.87 to 201.34] — luspatercept - placebo

19. Secondary Outcome: Post-Baseline Transfusion Event Frequency
Description: The number of transfusion events after start of study treatment were evaluated. For the definition of transfusion events, if multiple transfusions happen on the same date, they are counted as one event; if multiple transfusions happen on two consecutive dates, they are counted as one event; if multiple transfusions happen on three consecutive dates, they are counted as two events. Results are presented in 24-week intervals, up to 96 weeks after start of study treatment
Time Frame: From first dose through 3 weeks post last dose (up to approximately 218 weeks)
Population: All randomized participants who received transfusions
Measure: Mean (Standard Deviation); unit: Number of transfusions
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 210 | 102
Number of transfusions
  Week 1 - 24 | 7.1 (2.03) | 7.9 (1.65)
  Week 25 - 48: number analyzed (Participants) | 201 | 96
  Week 25 - 48 | 7.0 (2.02) | 7.6 (1.61)
  Week 49 - 72: number analyzed (Participants) | 177 | 62
  Week 49 - 72 | 7.0 (2.04) | 7.5 (1.28)
  Week 73 - 96: number analyzed (Participants) | 155 | 3
  Week 73 - 96 | 7.0 (2.13) | 7.0 (1.00)

20. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Apparent Clearance (CL/F)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
L/day | 0.437 (38.5) |

21. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Apparent Volume of Distribution of the Central Compartment (V1/F)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
Liters | 7.08 (26.7) |

22. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Elimination Half-life (t1/2)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
days | 11.2 (25.7) |

23. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Time to Reach Maximum Concentration (Tmax)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
Days | 5.48 [3.35 to 7.74] |

24. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Maximum Concentration for the Starting Dose (Cmax)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
μg/mL | 5.64 (25.1) |

25. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Maximum Concentration at Steady State for the Starting Dose (Cmax,ss)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
μg/mL | 8.31 (30.1) |

26. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Area Under the Concentration-Time Curve at Steady State for the Starting Dose (AUCss)
Time Frame: Blood serum samples taken pre-dose and on Days 1, 22, 64, 85, 106, 127, 169, 211, 253, 295, 337
Population: All randomized participants with available PK measurements for Luspatercept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 0
day*μg/mL | 129 (36.0) |

27. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. A serious AE is any AE occurring at any dose that - Results in death - Is life-threatening - Requires or prolongs existing inpatient hospitalization - Results in persistent or significant disability/incapacity - Is a congenital anomaly/birth defect - Constitutes an important medical event. The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03): - Grade 1 = Mild - Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention) - Grade 3 = Severe (limitation in activity; medical intervention required) - Grade 4 = Life-threatening - Grade 5 = Death
Time Frame: From first dose to 90 days following last dose (up to approximately 52 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 223 | 109
Participants
  ≥ 1 Treatment-emergent adverse event (TEAE) | 219 | 102
  Serious TEAE | 53 | 8
  Grade ≥ 3 TEAE | 84 | 19
  Treatment-related TEAE | 135 | 31
  Treatment-related Serious TEAE | 13 | 0
  Treatment-related TEAE ≥ Grade 3 | 27 | 1
  TEAE leading to death | 2 | 1
  Trt-related TEAE leading to death | 0 | 0
  TEAE leading to dose reduction | 10 | 3
  TEAE leading to dose delay | 46 | 11
  TEAE leading to drug discontinuation | 25 | 2
  Trt-related TEAE leading to dose reduction | 9 | 2
  Trt-related TEAE leading to dose delay | 15 | 3
  Trt-related TEAE leading to drug discontinuation | 20 | 1

28. Secondary Outcome: Participants With Pre-Existing and/or Treatment-Emergent Antidrug Antibodies (ADA)
Description: Number of participants with positive ADA prior to taking study drug and/or during study. A participant was counted as "treatment-emergent" if there was a positive post-baseline sample while the baseline sample was ADA negative, or there was a positive post-baseline sample with a titer ≥ 4-fold of the baseline titer while the baseline sample was ADA positive. A participant was counted as "preexisting" if the baseline sample was ADA positive and the participant was not qualified for "treatment-emergent."
Time Frame: Timeframe: pre-dose, Day 1, Days 22, 64, 106, 148, 232, 316
Population: All treated participants with available measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept + BSC | Placebo + BSC
Number analyzed (Participants) | 221 | 109
Participants
  Pre-existing | 2 | 1
  Treatment-emergent | 4 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (approximately 56 months) SAEs and NSAEs were assessed from first dose to 90 days following last dose (up to approximately 52 months)
Description: Adverse events were collected in all participants who received at least 1 dose of study drug.
Arm/Group | Luspatercept + BSC | Placebo + BSC
All-Cause Mortality (participants affected / at risk) | 4/223 | 1/109
Serious Adverse Events (participants affected / at risk) | 53/223 | 8/109
Other Adverse Events (participants affected / at risk) | 211/223 | 95/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept + BSC (N=223) | Placebo + BSC (N=109)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac iron overload (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0
Dengue fever (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Parotid abscess (Infections and infestations) | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 0
Splenic abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral sepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Coombs direct test positive (Investigations) | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute erythroid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept + BSC (N=223) | Placebo + BSC (N=109)
Abdominal pain (Gastrointestinal disorders) | 30 | 7
Abdominal pain upper (Gastrointestinal disorders) | 25 | 8
Constipation (Gastrointestinal disorders) | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 41 | 14
Dyspepsia (Gastrointestinal disorders) | 19 | 1
Nausea (Gastrointestinal disorders) | 29 | 6
Toothache (Gastrointestinal disorders) | 15 | 5
Vomiting (Gastrointestinal disorders) | 30 | 8
Asthenia (General disorders) | 26 | 11
Fatigue (General disorders) | 38 | 16
Influenza like illness (General disorders) | 21 | 8
Injection site pain (General disorders) | 12 | 3
Pain (General disorders) | 14 | 4
Pyrexia (General disorders) | 47 | 24
Gastroenteritis (Infections and infestations) | 18 | 9
Influenza (Infections and infestations) | 25 | 8
Nasopharyngitis (Infections and infestations) | 17 | 4
Pharyngitis (Infections and infestations) | 36 | 15
Tonsillitis (Infections and infestations) | 16 | 2
Upper respiratory tract infection (Infections and infestations) | 93 | 43
Urinary tract infection (Infections and infestations) | 13 | 6
Fall (Injury, poisoning and procedural complications) | 8 | 8
Transfusion reaction (Injury, poisoning and procedural complications) | 12 | 5
Alanine aminotransferase increased (Investigations) | 12 | 4
Liver iron concentration increased (Investigations) | 12 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 16 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 72 | 33
Bone pain (Musculoskeletal and connective tissue disorders) | 50 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 14 | 9
Osteoporosis (Musculoskeletal and connective tissue disorders) | 13 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 12
Spinal pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Dizziness (Nervous system disorders) | 29 | 5
Headache (Nervous system disorders) | 78 | 27
Lethargy (Nervous system disorders) | 12 | 4
Menstruation irregular (Reproductive system and breast disorders) | 12 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 41 | 13
Urticaria (Skin and subcutaneous tissue disorders) | 17 | 4
Hypertension (Vascular disorders) | 23 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT02604433/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT02604433/SAP_002.pdf